CLINICAL TRIAL: NCT06601322
Title: Functional Outcomes in CondUction System Pacing and Right Ventricular Synchrony The FOCUS-Right Pilot Study (FOCUS-Right)
Brief Title: Functional Outcomes in CondUction System Pacing and Right Ventricular Synchrony (FOCUS-Right)
Acronym: FOCUS-Right
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20028599
Record Dates: First submitted 2024-07-09; First posted 2024-09-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Left Branch Bundle Block; RV - Right Ventricular Abnormality
Keywords: Pacemaker; CPET-CMR
MeSH Terms: conditions — Bundle-Branch Block | interventions — epicatechin gallate; Exercise Test; Clostridium perfringens epsilon-toxin

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized controlled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Ventricular Pacing (NVP) (Other): Assessment 1 (No Ventricular Pacing) will be performed with no ventricular pacing to assess baseline right and left ventricular function at rest and during exercise.
  Interventions: Other: Pacemaker Interrogation and Electrocardiogram (ECG):; Other: Cardiopulmonary Exercise Test (CPET) and Exercise Stress Cardiac Magnetic Resonance (ExeCMR; Other: Continuous pacemaker telemetry (CPT)
- Non-selective or Selective Left Bundle Branch Area Pacing (nsLBBAP) (Active Comparator): Phase 2 (non-selective or selective Left Bundle Branch Area Pacing or ns/sLBBAP) will assess right and left ventricular function at rest and during exercise with non-selective or selective left bundle branch area pacing
  Interventions: Other: Pacemaker Interrogation and Electrocardiogram (ECG):; Other: Cardiopulmonary Exercise Test (CPET) and Exercise Stress Cardiac Magnetic Resonance (ExeCMR; Other: Continuous pacemaker telemetry (CPT)
- Left Bundle Branch Area Pacing with Anodal Capture (aLBBAP) (Experimental): Phase 3 (Left Bundle Branch Area Pacing with Anodal Capture or aLBBAP) will assess right and left ventricular function at rest and during exercise with left bundle branch area pacing with anodal capture.
  Interventions: Other: Pacemaker Interrogation and Electrocardiogram (ECG):; Other: Cardiopulmonary Exercise Test (CPET) and Exercise Stress Cardiac Magnetic Resonance (ExeCMR; Other: Continuous pacemaker telemetry (CPT)

INTERVENTIONS:
Other: Pacemaker Interrogation and Electrocardiogram (ECG): — Prior to the CMR study, subjects will undergo baseline interrogation of their dual chamber LBBAP to assess for appropriate device function. Lead capture characteristics will then be assessed with continuous intracardiac electrogram characteristics recorded from the atrial and ventricular lead with simultaneous 12-lead ECG rhythm strip recordings to assess for settings at which the investigators can differentiate aLBBAP, sLBBAP and nsLBBAP. Pacing output will be increased until left bundle branch area pacing with anodal capture is achieved, and then decreased until anodal capture is lost. These programming parameters will be recorded and utilized for Phase 2-3 of the CPET-CMR scan. 12-lead ECG rhythm strips of QRS morphology with each parameter set will be obtained and saved for later analysis.
Other: Cardiopulmonary Exercise Test (CPET) and Exercise Stress Cardiac Magnetic Resonance (ExeCMR — Following ECG and pacemaker analysis as above for safety, subjects will be fitted with 2 sets of MRI-compatible ECG monitoring systems a BP monitoring system , and a finger-tip pulse gating system. Imaging will be performed on a Magnetom Vida 3 Tesla scanner by trained CRM radiology technologists.
Other: Continuous pacemaker telemetry (CPT) — CPT will be established and supervised by a cardiac electrophysiologist to monitor for evidence of noise or artifact which may lead to inability to appropriately sense native atrial depolarization in DDD mode. Subjects with PM dependence are excluded. If noise is noted during scanning with NVP, then scanning will NOT be performed during P-synchronous pacing and will instead be performed during overdrive pacing at a rate above the patients maximal achieved heart rate with exertion during Phase 1. Thus, there is minimal risk to the subject from PM programming during CPET-CMR.

SUMMARY:
The goal of this prospective single center clinical trial is to evaluate the safety and feasibility of performing simultaneous exercise stress cardiac magnetic resonance (CPET-CMR) and cardiopulmonary exercise testing in patients with pre-existing left bundle branch area pacemakers (LBBAP) programmed to an atrial sensing mode. Measurements of right ventricular, left ventricular function, and exercise capacity will be obtained at various LBBAP programming parameters at rest and during low intensity exercise. The main aims of the study are:

* Demonstrate the safety and feasibility of performing CPET-CMR in patients with pre-existing LBBAP programmed to P-synchronous ventricular pacing mode.
* Generate preliminary data evaluating differences in RV function, LV function, and exercise capacity during various pacemaker programming settings.

DETAILED DESCRIPTION:
Conduction system pacing, namely left bundle branch area pacing (LBBAP) represents an important pacing modality introduced to avoid the deleterious effects of non-physiologic ventricular activation during chronic right ventricular pacing and /or left bundle branch block (LBBBP). Previous studies have demonstrated that LBBAP exhibits similar or superior left ventricular resynchronization compared to conventional treatment modalities, the impact of this novel pacing strategy on the right ventricle has not yet been addressed. This study aims to demonstrate the safety and feasibility of assessing LBBAP performance with a focus on right ventricular function in a novel way utilizing Cardiopulmonary Exercise Testing and Exercise Stress Cardiac Magnetic Resonance.

The investigators plan a 1-day prospective non-randomized controlled pilot study in which up to 20 subjects with left bundle branch area pacemakers with evidence of output dependent anodal capture will undergo low intensity exercise CPET-CMR at three different LBBAP settings (underlying rhythm, non-selective left bundle pacing, non-selective left bundle pacing with anodal stimulation).

ELIGIBILITY:
Inclusion Criteria:

* presence of dual chamber LBBAP implantation
* presence of anodal capture with bipolar pacing configuration as determined at pacing implant.

Exclusion Criteria:

* Known history of chronotropic incompetence
* high degree or complete heart block
* inability to tolerate NVP during initial device interrogation
* pregnancy
* inability to undergo MRI or exercise utilizing supine bicycle at target work-load
* presence of MRI unsafe pacemaker components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pacemaker Atrial (P Wave) Over-Sensed Events | Day 1: From beginning of CPET-CMR imaging procedure to end of CPET-CMR imaging procedure on study day.
  Incidence of pacemaker atrial (P Wave) over sensing as derived from continuous pacemaker telemetry at optimal programmed atrial sensitivity.

SECONDARY OUTCOMES:
Incidence of Pacemaker Atrial (P Wave) Under-Sensed Events | Day 1: From beginning of CPET-CMR imaging procedure to end of CPET-CMR imaging procedure on study day.
  Incidence of pacemaker atrial (P Wave) under sensing as derived from continuous pacemaker telemetry at optimal programmed atrial sensitivity.
Left Ventricular Ejection Fraction (%) | Day 1: From beginning of CPET-CMR imaging procedure to end of CPET-CMR imaging procedure on study day.
  Left ventricular ejection fraction (%) as measured by cardiac magnetic resonance imaging.
Right Ventricular Ejection Fraction (%) | Day 1: From beginning of CPET-CMR imaging procedure to end of CPET-CMR imaging procedure on study day.
  Right ventricular ejection fraction (%) as measured by cardiac magnetic resonance imaging.

OTHER OUTCOMES:
Slope of VO2 as a Function of Work Rate | Day 1: From beginning of CPET-CMR imaging procedure to end of CPET-CMR imaging procedure on study day.
  Slope of VO2 as a function of work rate as quantified by cardiopulmonary exercise testing.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Pillai, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No